CLINICAL TRIAL: NCT04440943
Title: A Phase 1 Study of the PD-L1xCD27 Bispecific Antibody CDX-527 in Patients With Advanced Malignancies
Brief Title: A Study of the PD-L1xCD27 Bispecific Antibody CDX-527 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX527-01
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer; Breast Cancer; Gastric Cancer; Renal Cell Carcinoma; Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Cholangiocarcinoma; Bladder Urothelial Carcinoma; MSI-H Colorectal Cancer; Esophageal Cancer; Hepatic Cancer; Head and Neck Cancer; Other Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Renal Cell; Ovarian Neoplasms; Fallopian Tube Neoplasms; Cholangiocarcinoma; Esophageal Neoplasms; Liver Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDX-527 (Experimental): Dose-escalation phase: Eligible patients will receive CDX-527 treatment based on cohort assigned until progression or intolerance.
  Expansion phase: Patients will receive CDX-527 at the dose level(s) chosen during the escalation phase.
  Interventions: Drug: CDX-527

INTERVENTIONS:
Drug: CDX-527 — CDX-527 is administered by infusion every 2 weeks

SUMMARY:
This is an open-label, non-randomized, multicenter, dose-escalation and expansion study in patients with selected solid tumors.

DETAILED DESCRIPTION:
This study will determine the safety, tolerability and activity of CDX-527.

Eligible patients that enroll to the dose-escalation portion of the study will be assigned to one of several dose levels of CDX-527. The dose-escalation part of the study will determine the safety profile of CDX-527 and determine which dose(s) of CDX-527 will be studied in the expansion part of the study.

The expansion part of the study will enroll eligible patients with certain solid tumors to be treated at dose(s) identified during dose-escalation

Up to 40 patients will be enrolled. All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Key Inclusion Criteria:

1. Recurrent, locally advanced or metastatic solid tumor cancer excluding the following: MSI-low colorectal cancer, glioblastoma multiforme, prostate cancer, pancreatic cancer, mucosal and ocular melanoma.
2. Receipt of all standard therapies for the tumor type
3. Measurable (target) disease by iRECIST
4. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 3 months following last treatment
5. Willingness to undergo a pre-treatment and on-treatment biopsy, if required

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other monoclonal antibodies.
2. Previous treatment with any anti-CD27 antibody.
3. Inadequate washout period from prior therapy as defined in the Protocol.
4. Patients who have received more than 0 or 1 prior PD-1/PD-L1 inhibitor depending on their tumor type
5. Major surgery within 4 weeks prior to study treatment.
6. Use of immunosuppressive medications within 4 weeks or systemic corticosteroids within 2 weeks prior to study treatment.
7. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers. For all other cancers, the patient must be disease-free for at least 3 years to be allowed to enroll.
8. Thrombotic events within the last 6 months prior to study treatment
9. Active, untreated central nervous system metastases.
10. Active autoimmune disease or documented history of autoimmune disease.
11. History of (non-infectious) pneumonitis or has current pneumonitis.
12. Active diverticulitis
13. Known infection of HIV, Hepatitis B, or Hepatitis C.

There are additional criteria your study doctor will review with you to confirm your eligibility for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of CDX-527 as assessed by CTCAE v5.0 | From first dose through 28 days after last dose
  The rates of drug-related adverse events will be summarized and maximum tolerated dose will be determined.

SECONDARY OUTCOMES:
Objective Response Rate | Every 8 weeks starting with first dose until disease progression, assessed up to approximately 1-2 years.
  The percentage of patients who achieve a confirmed immune complete response (iCR) or immune partial response (iPR)
Clinical Benefit Rate | Every 8 weeks, starting with first dose until disease progression, assessed up to approximately 1-2 years.
  The percentage of patients who achieve best response of confirmed iCR or iPR, or immune stable disease (iSD) for at least four months
Duration of Response | First occurrence of a documented objective response to disease progression or death (up to approximately 1-2 years)
  The interval from which measurement criteria are first met for iCR or iPR until the first date that progressive disease is objectively documented
Progression-free Survival | From the first dose to the first occurrence of disease progression or death due to any cause (up to approximately 1-2 years)
  The time from start of study drug to time of progression or death, whichever occurs first
Overall Survival | The time from start of study drug to death from any cause (up to approximately 1-2 years)
  The time from start of study drug to death
Immunogenicity Evaluation | Prior to the first dose of study treatment, then intermittently before dosing, and up to 60 days after the last dose
  Serum samples will be obtained for assessment of human anti-CDX-527 antibodies
Pharmacokinetic Evaluation | Before and after dosing, with additional timepoints after the first two doses, then intermittently before dosing and up to 60 days after the last dose
  CDX-527 serum concentrations will be measured at specified visits.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northside Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Duke Cancer Center, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon